CLINICAL TRIAL: NCT07270458
Title: Clinical Evaluation of Pain Perception and Patient Acceptance During Chemomechanical Caries Removal Using Cariclast Versus Conventional Caries Removal in 2nd Primary Molars With Occlusal Caries in Children: A Randomized Clinical Trial
Brief Title: Clinical Comparison of Cariclast Gel and Rotary Drilling Technique for Caries Removal in 2d Primary Molars
Acronym: CARICLAST-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noran Mohamed Kamel Bayoumi, Nora mohamed kamel, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK2025-CARICLAST
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries in Primary Molars
Keywords: Chemomechanical caries removal; Rotary method; Sodium hypochlorite gel; caries removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cariclast group (Experimental): Participants in this arm will undergo chemomechanical caries removal using Cariclast gel (sodium hypochlorite-based CMCR agent). The gel will be applied on the carious lesion according to the manufacturer's instructions, followed by gentle removal of the softened dentin using hand excavators.
  Interventions: Procedure: cares removal using cariclast gel
- Conventional Mechanical Caries Removal (Active Comparator): Participants in this arm will undergo conventional mechanical caries removal using a high-speed rotary handpiece under adequate water cooling. The procedure will follow standard clinical principles for removing infected dentin while maintaining a conservative approach to preserve sound tooth structure in primary molars.
  Interventions: Procedure: Conventional Mechanical Caries Removal

INTERVENTIONS:
Procedure: cares removal using cariclast gel — Chemomechanical caries removal using Cariclast gel applied to soften infected dentin, followed by gentle excavation with hand instruments.
  Other Names: Sodium hypochlorite-based CMCR agent
  Arms: cariclast group
Procedure: Conventional Mechanical Caries Removal — Conventional mechanical caries removal performed using a high-speed rotary handpiece under adequate water cooling, following standard clinical principles for primary molars.
  Arms: Conventional Mechanical Caries Removal

SUMMARY:
This randomized clinical trial aims to compare two different methods of caries removal in primary molars: the chemomechanical technique using Cariclast gel and the conventional rotary drilling method. The study will evaluate and compare the pain perception, patient acceptance, and operative time associated with both techniques in children aged 5-7years.

DETAILED DESCRIPTION:
Dental caries is one of the most common chronic diseases in children, and the management of carious lesions in primary teeth should be both effective and minimally invasive. Traditional caries removal using rotary instruments is associated with discomfort and anxiety among pediatric patients.

Chemomechanical caries removal (CMCR) agents such as Cariclast have been developed as a more conservative and less traumatic alternative. Cariclast works by softening the infected dentin chemically, allowing its gentle removal without pain or vibration.

This randomized controlled clinical trial will compare Cariclast with the conventional rotary drilling method regarding:

Pain perception assessed using the FLACC scale.

Patient acceptance evaluated using the Visual Analog Scale (VAS).

Operative time required to complete the caries removal procedure.

All procedures will be performed on cooperative children with occlusal caries in primary molars, without pulpal involvement, attending the Pediatric Dentistry Department, Faculty of Dentistry, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* Children:

  1. children aged 4-7 years
  2. in good general health, and medically free according to parent history.
  3. Cooperative patients
  4. Children whom their parents will comply with follow-ups.
  5. Children whom their parents who accept to sign informed consent

Tooth:

1. Broad cavitated occlusal lesion with dentinal involvement
2. (Black's Class I cavity) and occlusal access.
3. Radiograph showing dentinal caries up to two-thirds of the dentinal thickness.
4. The consistency of carious lesions ranges from soft to medium hard.
5. Color of carious lesion ranges from light yellow to brown

Exclusion Criteria:

* Children:

  1. Medically or developmentally compromising conditions
  2. Children who will be unable to attend follow-up visits.
  3. Children whom their parents refuse to give written formed consent.

Teeth:

1. Cases requiring restorative treatment that is not of the Class I variety.
2. Extensively damaged teeth.
3. Radiograph showing dentinal caries of more than two thirds of the dentinal thickness.
4. Caries involving pulp or extending below the gingiva.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain Perception During Caries Removal | During the caries removal procedure (immediate intraoperative assessment)
  Pain perception will be evaluated using the Wong-Baker FACES Pain Rating Scale. Before starting caries removal, the child will be briefly shown the six facial expressions and given age-appropriate instructions to ensure proper understanding of how to express discomfort. During the procedure, immediately at the moment of peak stimulation, the child will be asked to point to the face that best reflects their pain experience. The selected score (ranging from 0 to 10) will be recorded as an objective standardized measure of procedural pain.

SECONDARY OUTCOMES:
Child Acceptance of the Caries Removal Technique | Immediately after the procedure
  Patient acceptance will be measured immediately after completion of the caries removal procedure using a Visual Analog Scale (VAS). The scale consists of a 100-mm horizontal line with descriptors at each end indicating the extremes of comfort, ranging from "no discomfort" to "worst possible discomfort." Each child will be asked to mark a point on the line that best represents their overall comfort during the procedure. The distance in millimeters from the "no discomfort" anchor to the child's mark will be measured to quantify the level of acceptance. Higher scores indicate lower acceptance of the technique.

CONTACTS AND LOCATIONS:
Overall Officials: randa youssef abdelgawad, professor, Study Director — Cairo University; rana sobhy saeed, Study Director — Cairo University

REFERENCES:
- [Result] Gupta N, Marwah N, Nigam A, Vishwanathaiah S, Alessa N, Almeslet A, Alhakami K, Dawood T, Masha FM, Maganur PC. Evaluation of Papacarie(R), Carie-Care, BRIX3000 and conventional hand instrumentation for caries removal in primary teeth: a randomized control study. J Clin Pediatr Dent. 2024 May;48(3):131-138. doi: 10.22514/jocpd.2024.066. Epub 2024 May 3. PMID 38755991
- [Result] Nagaveni, N. B., Radhika, N. B., Satisha, T. S., Ashwini, K. S., Sridhar, N., & Gupta, S. (2016). Efficacy of new chemomechanical caries removal agent compared with conventional method in primary teeth: An in vivo study. International Journal of Oral Health Sciences, 6(2), 52-58. doi: 10.4103/2231-6027.199986
- [Result] Cardoso M, Coelho A, Lima R, Amaro I, Paula A, Marto CM, Sousa J, Spagnuolo G, Marques Ferreira M, Carrilho E. Efficacy and Patient's Acceptance of Alternative Methods for Caries Removal-a Systematic Review. J Clin Med. 2020 Oct 23;9(11):3407. doi: 10.3390/jcm9113407. PMID 33114249
- [Result] Al Agili DE. A systematic review of population-based dental caries studies among children in Saudi Arabia. Saudi Dent J. 2013 Jan;25(1):3-11. doi: 10.1016/j.sdentj.2012.10.002. Epub 2012 Nov 10. PMID 23960549
- [Result] Chaussain-Miller C, Decup F, Domejean-Orliaguet S, Gillet D, Guigand M, Kaleka R, Laboux O, Lafont J, Medioni E, Serfaty R, Toumelin-Chemla F, Tubiana J, Lasfargues JJ. Clinical evaluation of the Carisolv chemomechanical caries removal technique according to the site/stage concept, a revised caries classification system. Clin Oral Investig. 2003 Mar;7(1):32-7. doi: 10.1007/s00784-003-0196-5. Epub 2003 Feb 20. PMID 12673435
- [Result] Kotb RM, Abdella AA, El Kateb MA, Ahmed AM. Clinical evaluation of Papacarie in primary teeth. J Clin Pediatr Dent. 2009 Winter;34(2):117-23. doi: 10.17796/jcpd.34.2.f312p36g18463716. PMID 20297701